CLINICAL TRIAL: NCT02401971
Title: Irinotecan Plus Thalidomide in Second Line Advanced Gastric Cancer : A Multicenter, Randomized, Controlled and Prospective Trial
Brief Title: Irinotecan Plus Thalidomide in Second Line Advanced Gastric Cancer
Acronym: ITAGC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wang Jufeng (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Henan Provincial People's Hospital (Other); Second Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Wang Jufeng, Master, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DREAM-002
Record Dates: First submitted 2015-02-25; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2014-09

CONDITIONS: Gastric Cancer
Keywords: Thalidomide; Irinotecan; Second Line
MeSH Terms: conditions — Stomach Neoplasms | interventions — Thalidomide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (thalidomide+CPT-11) (Experimental): Patients will receive CPT-11 180 mg/m^2 ivgtt ,over 90 minutes on day 1, every 21 days for one cycle, four cycles ,and oral thalidomide 100 mg/d qn. Maintenance therapy with thalidomide in the same dose is performed until disease progression.
  Interventions: Drug: Thalidomide; Drug: CPT-11
- Arm B (CPT-11) (Experimental): Patients will receive CPT-11 180 mg/m^2 ivgtt ,over 90 minutes on day 1, every 21 days for one cycle, four cycles.
  Interventions: Drug: CPT-11

INTERVENTIONS:
Drug: Thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid
  Arms: Arm A (thalidomide+CPT-11)
Drug: CPT-11 — Given Ivgtt
  Other Names: Irinotecan hydrochloride; Campto; Camptosar; irinotecan; U-101440E

SUMMARY:
Recent clinical studies have demonstrated a reduction of irinotecan (CPT-11) gastrointestinal toxicities when the CPT-11 is administered in combination with thalidomide in patients with diagnosis of gastric cancer. The main purpose of this study is to investigate the efficacy and safety of thalidomide and CPT-11 in advanced gastric cancer. The investigators will also manage to find out the possible interactions between CPT-11 pharmacokinetics and thalidomide to explain the previously described gastrointestinal toxicity reduction.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center, controlled clinical trial, aimed to evaluate efficacy and tolerability of thalidomide and CPT-11 in advanced gastric cancer. A total of 900 patients are planned to be enrolled into the study. Patients with diagnosis of advanced gastric cancer will be randomized into two groups, and be treated with thalidomide+ CPT-11 or CPT-11, respectively. The primary end point is time to progression (TTP), and the secondary end points include efficacy, overall survival (OS) and the occurrence of delayed diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* 18y <Age<75y
* Patients with histologically proven tumor focus will be eligible for this protocol
* Measurable or assessable disease
* At least 4 weeks since last chemotherapy ;chemotherapy regimens without Irinotecan
* No hepatic, renal and hematopoietic dysfunction; no hemorrhage of digestive tract,obstructive jaundice, gastrointestinal perforation or obstruction
* ECOG PS:0-2
* Expected OS ≥ 3 months

Exclusion Criteria:

* obstruction of digestive tract, thrombosis or other intolerant side effects during treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
time to progression(TTP) | up to 2 months

SECONDARY OUTCOMES:
complete response rate (CRR) for advanced gastric cancer | up to 2 months
overall survival (OS) | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jufeng, Study Chair — Henan Cancer Hospital; Qin Yanru, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Zhou Yun, Principal Investigator — Henan Provincial People's Hospital; Zhang Zhongmian, Principal Investigator — Second Affiliated Hospital of Zhengzhou University; Guo Yanzhen, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China